CLINICAL TRIAL: NCT01569256
Title: The Effect Of Cabergoline On Follicular Microenvironment Profile In Patients With High Risk Of Ohss
Brief Title: Ovarian Hyperstimulation Syndrome and Cabergoline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etlik Zubeyde Hanim Womens' Health and Teaching Hospital (Unknown)
Responsible Party: Principal Investigator, Assoc. Prof. Emine Seda Guvendag Guven, Assoc. Prof., Etlik Zubeyde Hanim Womens' Health and Teaching Hospital
Organization: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ESG1
Record Dates: First submitted 2012-03-26; First posted 2012-04-03 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Polycystic Ovarian Syndrome; Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome | interventions — Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabergoline administered group (Active Comparator): The patients in this group will have cabergoline (Dostinex tablet, Pfizer, Istanbul, Turkey, started on day of HCG, 0.5 mg/day for 8 days) for prevention of OHSS.
  All patients were administered long luteal protocol for ovulation induction.
  Interventions: Drug: Cabergoline
- Control arm (No Intervention): The patients in the control group had no manipulation for prevention of OHSS and age-, BMI-matched with the active comparator group.
  All patients were administered long luteal protocol for ovulation induction.

INTERVENTIONS:
Drug: Cabergoline — Cabergoline tablet, Pfizer, Istanbul, Turkey, started on day of HCG, 0.5 mg/day for 8 days
  Other Names: Dostinex
  Arms: Cabergoline administered group

SUMMARY:
Cabergoline prevents ovarian hyperstimulation syndrome in high risk patients by disrupting follicular fluid hormone microenvironmentally altering the follicular fluid levels of insulin like growth hormone -I (IGF-I), antimullerian hormone (AMH), inhibin B and hepatocyte growth factor (HGF) levels in women with PCOS and high risk of ovarian hyperstimulation syndrome (OHSS).

DETAILED DESCRIPTION:
Dopamine agonists have been proposed as a prophylactic treatment for OHSS in women with high risk of OHSS, however the possible mechanism of action has not been clearly known. In experimental studies, inhibition of vascular endothelial growth factor based pathway was proposed as a possible action of mechanism of dopamine agonists. However the role hepatocyte growth factor (HGF), insulin like growth factor-I (IGF-I), inhibin B and antimullerian hormone (AMH) on cabergoline action in OHSS prevention has not been known.

ELIGIBILITY:
Inclusion Criteria:

* Development of more than 14 leading follicles larger than 10 mm and serum estradiol more than 3000 pg/ml at the end of ovulation induction with long luteal ovulation induction protocol.
* Having the criteria of PCOS

Exclusion Criteria:

* Not having the inclusion criteria.

Ages: 23 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Concentrations of follicular fluid AMH | 1 year

SECONDARY OUTCOMES:
Concentrations of follicular fluid inhibin B | 1 year
Concentrations of follicular fluid HGF | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Emine Seda Guvendag Guven, MD, Study Chair — Rize University, Faculty of Medicine